CLINICAL TRIAL: NCT02067312
Title: Effects of Traditional Thai Massage on Pain and Pain Related Parameters in Patients With Upper Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Vitsarut Buttagat, Mae Fah Luang University, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55218152
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thai massage (Experimental): The participants will receive a thirty minutes session of Thai massage onto the trapezius muscle
  Interventions: Other: Thai massage
- Sham Microwave diathermy (Sham Comparator): The participants will receive a thirty minutes session of Sham microwave diathermy onto the trapezius muscle
  Interventions: Other: Thai massage

INTERVENTIONS:
Other: Thai massage

SUMMARY:
The purpose of this study is to determine the effect of Thai massage on pain related parameters including Pain intensity, 24 hours pain intensity, Pressure pain threshold, anxiety, muscle tension, cervical range of motion, pain frequency, patient satisfaction and side effect in patients with chronic upper back pain associated with myofascial trigger points

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 - 50 years old
* The participants have experienced spontaneous upper pain for longer than 12 weeks (chronic) and that at least one trigger point will be present in the s trapezius muscles. Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition.
* The participants will be able to follow instructions.
* Good communication and cooperation.

Exclusion Criteria:

* A history of the following diseases or disorders:
* Cervical radiculopathy
* Contraindications of traditional Thai massage
* Contagious skin disease
* Injury or inflammation of muscle
* Bone fracture and/or joint dislocation
* Open wound
* Uncontrolled hypertension
* Drug and/or alcohol intoxication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain score on Visual analog scale | 5 weeks
  The intensity of pain will be reported by the participant on a visual analog scale ranging from 0 to 10. Zero indicates no pain anywhere and 10 indicates the most pain ever experienced.

SECONDARY OUTCOMES:
Pressure Pain Threshold as a measure by algometry | 5 weeks
Muscle tension on Visual analog scale | 5 weeks
Anxiety on State Anxiety Inventory | 5 weeks
Cervical range of motion as a measure by Cervical Range of Motion Goniometer | 5 weeks
Pain intensity on McGill Pain Questionnaire | 5 weeks
Pain frequency occurred per week | 5 weeks
24 hours pain intensity on Visual analog scale | 5 weeks
Patient satisfaction level | 3 weeks
Number of Participants with Adverse Events | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Science, Mae Fah Luang University, Mueang, Changwat Chiang Rai, Thailand